CLINICAL TRIAL: NCT00195936
Title: Effect of Calcimimetic (Cinacalcet) on Phosphate-Induced Hyperparathyroidism in Children With Hypophosphatemic Rickets
Brief Title: Effect of Cinacalcet on Parathyroid Hormone Secretion in Children and Adolescents With Hypophosphatemic Rickets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05 02-027
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Hypophosphatemic Rickets, X-Linked Dominant
Keywords: Cinacalcet; PTH; XLH; children and adolescents with hypophosphatemic rickets (XLH)
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — Cinacalcet

ARMS (1):
- Overall Study (Experimental): Calcimimetics as an Adjuvant Treatment for Familial Hypophosphatemic Rickets
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet — Single oral dose of Cinacalcet for children with Hypophosphatemic Rickets

SUMMARY:
This study will measure the effect of cinacalcet (Sensipar) on parathyroid hormone (PTH) secretion in children and adolescents with hypophosphatemic rickets (XLH). The investigators are seeking evidence that patients with XLH may benefit from treatment with cinacalcet by achieving better control of PTH secretion.

DETAILED DESCRIPTION:
X-linked hypophosphatemic rickets (XLH) is an X-linked dominant genetic disorder. Common findings are low serum phosphate and inadequate 1,25(OH)2 vitamin D production. It is generally believed that the primary defect in XLH is impaired renal tubular transport of phosphate coupled with abnormal regulation of the enzyme responsible for the 1-alfa hydroxylation of 25(OH) vitamin D. The current treatment of children with XLH is large oral doses of phosphate and 1,25-dihydroxyvitamin D. There are two common side effects to this treatment; nephrocalcinosis and secondary hyperparathyroidism (HPT). The latter at times may cause hypertension, hypercalcemia, and permanent renal damage. The complication of secondary hyperparathyroidism is seen in 20% of the patients. The release of PTH from the glands into the circulation is tightly regulated by serum calcium concentration. The glands "read" serum calcium concentration via Ca sensing receptors (CaR) which are located at the surface of the glands. Calcimimetics are compounds that allosterically modulate the CaR, thereby enhancing its sensitivity to circulating serum calcium concentrations and consequently decreasing PTH secretion. When used in primary HPT, they rapidly reduce PTH level and normalize serum calcium concentration.

Cinacalcet is a calcimimetic agent recently approved by the FDA for treating hypercalcemia in patients with parathyroid carcinoma and secondary HPT in patients with chronic renal disease. Cinacalcet was found to be effective in decreasing both PTH level and the calcium X phosphorous ion product in dialysis patients.

The goal of our proposed acute study is to see whether concomitant administration of Cinacalcet and phosphate, to patients with XLH, will block completely or partially secretion of PTH (day 2), expected to be seen following administration of phosphate alone (day 1). We will also monitor serum phosphate, total calcium, and ionized calcium concentration to learn to what extent, if any, blockage of PTH secretion affects mineral homeostasis under this condition.

If found to be effective in blocking PTH secretion, Cinacalcet will become a candidate for a long-term study in children with XLH to protect them from developing secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Established patients with XLH
* Age 5 years old and above
* Normal serum calcium and creatinine concentrations

Exclusion Criteria:

* Patients with hypersensitivity to any component(s) of cinacalcet
* Hypocalcaemia
* Elevated serum creatinine

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change of serum Parathyroid Hormone (PTH) with use of cinacalcet | Baseline, 30 minutes, and 4 hours post dose

SECONDARY OUTCOMES:
Change of mineral homeostasis; ionized calcium, total calcium, and phosphate with use of calcimimetic | Baseline, 30 minutes, and 4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Levy-Olomucki, MD, Principal Investigator — Section of Pediatric Nephrology, Children's Mercy Hospitals and Clinics
Locations (1):
- Section of Pediatric Nephrology, Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States